CLINICAL TRIAL: NCT00104000
Title: The Effect of Surface Electrical Stimulation on Hyo-Laryngeal Movement in Healthy Individuals at Rest and During Swallow
Brief Title: Effect of Surface Electrical Stimulation on Movement of the Larynx
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050099; 05-N-0099
Record Dates: First submitted 2005-02-17; First posted 2005-02-18 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-01

CONDITIONS: Healthy
Keywords: Neuromuscular; Elevation; Current; Videofluoroscopy; Nasoendoscopy; Healthy Volunteer; HV

SUMMARY:
This study will examine whether surface electrical stimulation on the skin of the throat will: 1) move the larynx (voice box); 2) move the vocal folds in the larynx; and 3) cause less movement of the larynx when applied during swallowing. It is important that the larynx moves up and forward while swallowing so that food does not go into the airway. A device called VitalStim® (Registered Trademark), which provides electrical stimulation to the skin on the neck and under the chin, is widely used to treat people who have problems swallowing. This study will determine if VitalStim can move the voice box or the vocal folds in the larynx. This information is important for patients who have long-term problems raising or closing their larynxes when they swallow.

Healthy volunteers between 20 and 60 years of age may be eligible for this study. Candidates are screened with a medical history, physical examination, electrocardiogram, and nasoendoscopy. For the latter procedure, the inside of the subject's nose is sprayed with a decongestant, opening the nasal passages. A small flexible tube called a nasoendoscope is passed through the nose to the back of the throat. The scope allows observation of the larynx while the subject speaks, sings, whistles and makes prolonged vowel sounds.

Participants are familiarized with the VitalStim device before beginning the experimental procedures. The device consists of two sets of electrodes and a stimulation unit. The electrodes are placed on the neck and under the chin. Stimulation causes different sensations, according to the intensity level. They include "tingling/crawling," "vibrating" "warm/burning," and "grabbing." Subjects then undergo the following procedures:

* Nasoendoscopy with muscle stimulation: The inside of the nose is sprayed with a decongestant and the nasoendoscope is passed through one nostril to the back of the throat. Electrodes are placed on the throat area and under the chin. Stimulation is delivered 10 times at various places on the neck and under the chin while the subject sits quietly. This test shows if the vocal folds in the voice box move with surface electrical stimulation.
* Videofluoroscopy with muscle stimulation at rest and during swallowing: This is an x-ray study of the head and neck during swallowing and at rest to determine how stimulation affects the level of the voice box in the neck. Electrodes are placed under the chin and on the throat. The subject swallows 5 milliliters of barium, a contrast material that can be seen easily on x-ray. The x-ray machine is turned on for a few seconds at a time during each swallow of the barium and another 10 times while the subject is remaining still without swallowing.

DETAILED DESCRIPTION:
Objectives:

The purpose of the current study is to determine whether:

1. Surface electrical stimulation at rest using various electrode placements produces different hyo-laryngeal movements of in healthy adult humans.
2. One surface electrical stimulation array (placement 3b) reduces hyo-larynegeal movement in healthy humans during swallowing.

Study Population: healthy adults

Design: This study will employ a repeated measures design. Surface electrodes will be used to stimulate submental and laryngeal muscles either alone or in combination both at rest and during swallowing while using videofluoroscopy and nasolaryngoscopy to record hyo-laryngeal movement.

Outcome Measures: Kinematic analyses of hyo-laryngeal movements using image processing and marking from video-recordings will quantify movement with stimulation.

ELIGIBILITY:
INCLUSION CRITERIA:

The Healthy volunteers will be without cardiac, pulmonary, neurological, otolaryngological, psychiatric or speech, swallowing and hearing problems as determined by medical history and examination by a physician.

EXCLUSION CRITERIA:

* History of Rheumatic fever, mitral valve prolapse, or cardiac arrhythmias as determined by medical history, physical and EKG. A physician will auscultate for cardiac murmurs prior to any study to exclude volunteers who might be at risk for endocarditis. Subjects will have an EKG as part of the screening for participation in the study.
* Pregnancy will exclude women from participation because the study involves radiation exposure.
* None of the Healthy volunteers will have a reduction in the range of vocal fold movement during the nasoendoscopy that might suggest laryngeal paralysis or paresis, joint abnormality or neoplasm.
* Healthy Volunteers who have a cardiac demand pacemaker, dementia, exhibit non-stop vocalization, significant reflux due to use of a feeding tube, or drug toxicity will not be included for VitalStim, as these are contraindications to use of the device.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 47
Dates: Start 2005-02; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Lundy DS, Smith C, Colangelo L, Sullivan PA, Logemann JA, Lazarus CL, Newman LA, Murry T, Lombard L, Gaziano J. Aspiration: cause and implications. Otolaryngol Head Neck Surg. 1999 Apr;120(4):474-8. doi: 10.1053/hn.1999.v120.a91765. PMID 10187936
- [Background] Kahrilas PJ, Lin S, Rademaker AW, Logemann JA. Impaired deglutitive airway protection: a videofluoroscopic analysis of severity and mechanism. Gastroenterology. 1997 Nov;113(5):1457-64. doi: 10.1053/gast.1997.v113.pm9352847.
- [Background] ECRI Health Technology Assessment Group. Diagnosis and treatment of swallowing disorders (dysphagia) in acute-care stroke patients. Evid Rep Technol Assess (Summ). 1999 Mar;(8):1-6. No abstract available. PMID 11925971